CLINICAL TRIAL: NCT04121234
Title: Pidemiology, Outcomes and Risk Factors for Mortality in Critically-Ill Women Admitted to an Obstetric High Dependency Unit in a Resource-Limited Setting
Brief Title: Critically-Ill Women Admitted to an Obstetric High Dependency Unit in a Resource-Limited Setting
Status: Completed | Type: Observational
Sponsor: Doctors with Africa - CUAMM (Other)
Responsible Party: Principal Investigator, Claudia Marotta, MD, MPH, Doctors with Africa - CUAMM
Other Study IDs: 070919CUAMM
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Maternal Death
Keywords: High dependency unit; critical care; obstetric critical care; maternal mortality.
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure: " being admitted to HDU with a red code to OEWS" — High Dependency Unit, a set of predefined variables was assessed at hospital admission, HDU admission and at discharge from HDU with the aim to investigate epidemiology, clinical outcomes and risk factors for mortality in critically-ill parturients admitted to an obstetric HDU in a high volume, urban resource-limited maternity hospital

SUMMARY:
Sierra Leone faces the highest maternal mortality ratio in the world. Despite this extreme burden, the potential roles of obstetric critical care and high dependency units (HDUs) in this and other resource-limited settings remain scarcely explored. This study investigated epidemiology, clinical outcomes and risk factors for mortality in critically-ill parturients admitted to an obstetric HDU in a high volume, urban resource-limited maternity hospital.

DETAILED DESCRIPTION:
This is a retrospective observational study in women admitted to the HDU of Princess Christian Maternity Hospital (PCMH), Freetown, Sierra Leone, from 2nd October 2017 to 2nd October 2018. The study received ethical approval and waiver of informed consent from the Sierra Leone Ethics and Scientific Review Committee (18/12/18).

A set of predefined variables was assessed at hospital admission, HDU admission and at discharge from HDU. The primary data source was the HDU patient chart, with data crosschecked with the hospital patient charts and the HDU admission book for quality control purpose. Data of hospital deliveries, admissions and mortality were form the hospital register and the maternal mortality hospital database. Data were retrospectively collected by a study physician (CM) and included: patient demographics; admission date and source; main reason for admission in hospital; main reason for admission to the HDU (classified as: haemodynamic instability; sepsis; haemorrhage; acute renal failure; neurological impairment; respiratory distress; severe malaria; coagulopathy; other diagnoses). These are clinical diagnoses included in the hospital checklist to facilitate communication of referral to HDU and are thus based on the clinical assessment of the attending physician rather than on a strict research definitions.

Vital signs and treatments collected at admission included body temperature, heart rate, respiratory rate, neurological status according to the AVPU scale, systolic and diastolic blood pressure, transcutaneous saturation (SpO2). The ratio between SpO2 and fraction of inspired oxygen (SpO2/FiO2) was also measured. The obstetric modified early warning score (OEWS) was also calculated.

Specific treatments received at any point during HDU stay were extracted from the patient file and included: oxygen supplementation, use of vasopressors, blood transfusions, antibiotic therapy, activation of the magnesium protocol for eclamptic seizures prevention and hypotensive treatment protocol with hydralazine. Point of care laboratory parameters such as capillary lactates levels and haemoglobin were collected when available. Time from PCMH admission to HDU admission was calculated. Length of stay and patient outcomes (classified as death in HDU, discharge to ward, or transfer to other facility) were reported at discharge.

ELIGIBILITY:
Inclusion Criteria:

* All women admitted at HDU of the PCMH from the 2nd October 2017 to the 2nd October 2018.

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All women admitted at HDU of the PCMH from the 2nd October 2017 to the 2nd October 2018.
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Morality in HDU | one year
  The primary endpoint was the association between modifiable and non-modifiable factors and mortality during HDU stay. HDU death was defined as death during HDU stay, i.e. from referral to HDU to discharge from HDU.

SECONDARY OUTCOMES:
Hospital mortality | One year
  Hospital mortality was death during the whole hospital stay.
Lenght of stay | One year
  Time between the hdu admission and the hdu discharge, in days.
OEWS at the admission | one year
  coded as: red, yellow, green
reasons of admission | One Year
  classified as: haemodynamic instability; sepsis; haemorrhage; acute renal failure; neurological impairment; respiratory distress; severe malaria; coagulopathy; other diagnoses
Time of admission | One year
  Night/day and Working days/weeknd
Treatments received | One year
  oxygen supplementation (yes/no), use of vasopressors (yes/no), blood transfusions (yes/no), antibiotic therapy (yes/no), activation of the magnesium protocol for eclamptic seizures prevention (yes/no) and hypotensive treatment protocol with hydralazine during the stay (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Christian Maternity Hospital, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No